CLINICAL TRIAL: NCT03748043
Title: the Effectiveness of Lactoferrin in Treatment of Iron Deficiency Anemia in Children With Chronic Tonsillitis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Shimaa Abdallah Ahmed, principal investigator, South Valley University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 171984
Record Dates: First submitted 2018-11-18; First posted 2018-11-20 (Actual); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Iron-deficiency
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — Lactoferrin; teferrol

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- lactoferrin+ferric hydroxide polymaltose (Experimental): lactoferrin 100 mg /day plus ferric hydroxide polymaltose 6 mg /kilogram body wight for 3 months
  Interventions: Drug: Lactoferrin; Drug: Ferric Hydroxide Polymaltose
- ferric hydroxide polymaltose (Experimental): 6 mg /kilogram body wight of ferric hydroxide poly maltose per day for 3 months
  Interventions: Drug: Ferric Hydroxide Polymaltose

INTERVENTIONS:
Drug: Lactoferrin — lactoferrin 100 mg per day plus ferric hydroxide polymaltose 6 mg /kilogram of Elemental iron
  Other Names: (Pravotin sachets, Hygint, Egypt)
  Arms: lactoferrin+ferric hydroxide polymaltose
Drug: Ferric Hydroxide Polymaltose — group 2 will receive ferric hydroxide polymaltose 6 mg /kilogram of elemental iron
  Other Names: haemojet syrp

SUMMARY:
the investigators will compare the response to iron deficiency anemia to lactoferrin plus ferrous poly maltose versus ferrous poly maltose in Children With Chronic Tonsillitis

DETAILED DESCRIPTION:
Iron deficiency is frequently present with chronic inflammatory disease.(1) Iron deficiency anemia results from decreased body's iron content due to blood loss, poor dietary iron intake, malabsorption, or increased iron requirement. Immune activation drives a diversion of iron to storage sites, particularly the mononuclear phagocytes system in liver and spleen leads to poor hemoglobinization and anemia. Iron deficiency and immune activation lead to disturbances of iron homeostasis.(2) this trial will compare the response to iron deficiency anemia to lactoferrin plus ferrous poly maltose versus ferrous poly maltose in Children With Chronic Tonsillitis

ELIGIBILITY:
Inclusion Criteria:

* children 3-17 years old with chronic tonsillitis

Exclusion Criteria:

* no other causes of Iron Deficiency Anemia

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2019-02-21 (Actual); Primary Completion 2019-05-30 (Estimated); Study Completion 2019-05-30 (Estimated)

PRIMARY OUTCOMES:
Increase in blood hemoglobin | 1,3 months
  mean difference in hemoglobin level between pre treatment and post treatment. mean difference in hemoglobin level between pre treatment and post treatment.
Increase in serum ferritin | 3 months
  mean difference in ferritin level between pre treatment and post treatment.

CONTACTS AND LOCATIONS:
Overall Officials: shimaa Ahmed, MD, Study Chair — South Valley University
Locations (1):
- South Valley University, Qina, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cappellini MD, Comin-Colet J, de Francisco A, Dignass A, Doehner W, Lam CS, Macdougall IC, Rogler G, Camaschella C, Kadir R, Kassebaum NJ, Spahn DR, Taher AT, Musallam KM; IRON CORE Group. Iron deficiency across chronic inflammatory conditions: International expert opinion on definition, diagnosis, and management. Am J Hematol. 2017 Oct;92(10):1068-1078. doi: 10.1002/ajh.24820. Epub 2017 Jul 7. PMID 28612425
- [Result] Nairz M, Theurl I, Wolf D, Weiss G. Iron deficiency or anemia of inflammation? : Differential diagnosis and mechanisms of anemia of inflammation. Wien Med Wochenschr. 2016 Oct;166(13-14):411-423. doi: 10.1007/s10354-016-0505-7. Epub 2016 Aug 24. PMID 27557596